CLINICAL TRIAL: NCT06435208
Title: Impact of Subgingival Instrumentation on Psychological Distress and Mental Health Status in Bruxers With Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIYANKAPERIO2024
Record Dates: First submitted 2024-05-17; First posted 2024-05-30 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Periodontal Diseases; Bruxism; Periodontitis; Distress, Emotional
MeSH Terms: conditions — Periodontal Diseases; Bruxism; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PERIODONTITIS BRUXISM (Experimental): subgingival instrumentation will be done in all participants
  Interventions: Other: Subgingival instrumentation

INTERVENTIONS:
Other: Subgingival instrumentation — All the participants will undergo scaling and root planning with hand scalers, curettes and ultrasonic scaler.

SUMMARY:
Bruxism is a non-functional repetitive jaw-muscle activity characterized by grinding or clenching the teeth. Bruxism, characterized by the involuntary grinding or clenching of teeth, is a prevalent parafunctional habit affecting individuals of all ages. Stress, anxiety, and depression are the psychological factors most commonly associated with the presence of bruxism.

DETAILED DESCRIPTION:
Bruxism, characterized by the involuntary grinding or clenching of teeth, is a prevalent parafunctional habit affecting individuals of all ages. Although the etiology is not known exactly, it has been suggested that bruxism is a multifactorial disorder. Periodontitis, a prevalent inflammatory condition affecting the periodontium, has been linked to bruxism in several studies. The coexistence of bruxism and periodontitis poses unique challenges in clinical management of periodontitis. Also, as periodontitis became chronic, the occurrence of depression increased. Stress, anxiety, and depression are the psychological factors most commonly associated with the presence of bruxism. Therefore, this study aims to investigate impact of subgingival instrumentation on psychological distress and mental health status in bruxers with periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients
* Patient having periodontitis with bruxism
* Age between 30-50 years

Exclusion Criteria:

* History of mental health disorder
* History of systemic disease
* History of drugs having the potential impact on periodontal status like phenytoin, cyclosporin, calcium-channel blockers or antidepressant drugs
* Pregnant or lactating females

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Psychological distress | BASELINE,2 MONTHS ,3 MONTHS
  Assessment of psychological distress will be done by using Kessler Psychological distress(K10)
Mental Health Status | Baseline, 2 months, 3 months
  Assessment of mental health status will be done by using mental health inventory 38

SECONDARY OUTCOMES:
periodontal parameter | Baseline, 2 month, 3 month
  periodontal probing depth
periodontal inflammation | Baseline, 2 month, 3 month
  bleeding on probing

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Chandela, BDS, Principal Investigator — PGIDS , ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No